CLINICAL TRIAL: NCT07228858
Title: Uterine Scar Resection During Repeat Cesarean Delivery in a Simple Modification to Prevent Uterine Niche Formation: Results of a Randomized Controlled Trial
Brief Title: Uterine Scar Resection During Repeat Cesarean Delivery to Prevent Uterine Niche Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Latif Ahmed Alnezamy, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC9-2-2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Section Complications; Scar Niche; Scarred Uterus
Keywords: Repeated cesarean section; Uterine niche; Scar resection; Residual myometrial thickness; Randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Eligible women were randomized (1:1) using a computer-generated sequence in blocks of 10. Allocation was concealed in sequentially numbered, opaque, sealed envelopes opened by a trained nurse after consent. Obstetricians were informed of assignment, while participants , investigator, and ultrasound assessors remained blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- uterine scar resection (Active Comparator): During repeat cesarean section, the previous uterine cesarean section scar was resected.
  Interventions: Procedure: Repeated cesarean section with previous uterine cesarean section scar resection; Diagnostic Test: Saline-infusion Sonohysterography
- Non scar resection (Active Comparator): Standard repeat cesarean section without previous uterine cesarean section scar resection.
  Interventions: Procedure: Repeated cesarean section without uterine scar resection; Diagnostic Test: Saline-infusion Sonohysterography

INTERVENTIONS:
Procedure: Repeated cesarean section with previous uterine cesarean section scar resection — After creating the bladder flap, the uterus was incised 5 mm cranial to the scar and extended laterally 5 mm beyond its ends. After delivery of the newborn, a 1 cm segment of uterine wall (5 mm above and 5 mm below the scar) was excised. The incision edges were approximated with a central vertical mattress suture, followed by double-layer continuous myometrial closure including decidua with visceral peritoneum closure.
  Arms: uterine scar resection
Procedure: Repeated cesarean section without uterine scar resection — Standard repeat cesarean section without scar resection, followed by double-layer continuous myometrial closure including decidua with visceral peritoneum closure.
  Arms: Non scar resection
Diagnostic Test: Saline-infusion Sonohysterography — At 6 months postpartum, all participants are to be evaluated by a single blinded sonographer experienced in niche assessment. First, transvaginal ultrasound was performed to exclude pregnancy or pelvic pathology, followed by saline-infusion sonohysterography (2D, sagittal and coronal views). A niche is defined as ≥ 2 mm myometrial indentation at the scar site. Niche depth, length, width, and residual myometrial thickness are to be recorded.

SUMMARY:
The purpose of the study is to evaluate whether resection of the previous cesarean scar at repeat cesarean delivery reduces uterine niche formation and related morbidity without increasing operative risks.

DETAILED DESCRIPTION:
After eligibility and consenting, multigravida women with ≥1 prior cesarean section scheduled for repeat cesarean section at ≥28 weeks' gestation for any indication were randomized to

* Study group: During repeat cesarean section, the prior uterine scar was resected. After creating the bladder flap, the uterus was incised 5 mm cranial to the scar and extended laterally 5 mm beyond its ends. Following delivery, a 1 cm segment of uterine wall (5 mm above and below the scar) was excised. The incision edges were approximated with a central vertical mattress suture, followed by double-layer continuous myometrial closure (including decidua) and visceral peritoneum closure.
* Control group: Standard repeat cesarean section without scar resection, followed by identical double-layer and peritoneal closure.

All procedures were performed by obstetricians trained in the protocol. All women received standard preoperative antibiotics, 24-hour postoperative prophylaxis, and 10 units intramuscular oxytocin after delivery.

At 6 months postpartum, all participants will undergo transvaginal ultrasound and saline infusion sonohysterography performed by a blinded, experienced examiner. Sagittal and coronal views willl be obtained, and niche presence, depth, length, width, and residual myometrial thickness are to be recorded.

Obstetricians were informed of assignment, while participants and ultrasound assessor are blinded.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 prior cesarean section at ≥28 weeks' gestation.
* Undergoing repeat cesarean section for any indication.
* Provided informed consent and agreed to 6-month postpartum follow-up.
* Not planning pregnancy during follow-up.

Exclusion Criteria:

* Uterine fibroids, multiple gestation, chorioamnionitis, placenta previa, placental abruption, or preeclampsia/eclampsia.
* Hepatic or renal dysfunction, uncontrolled diabetes, or hemoglobin <10 g/dL.
* Systemic uncontrolled disease, chronic corticosteroid use, or smoking.
* Inability to provide informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2025-02-09 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of uterine niche formation after repeated cesarean section | At 6 months postpartum
  Using saline-infusion sonohysterography (2 dimensional, sagittal and coronal views). A niche is defined as ≥ 2 mm myometrial indentation at the scar site.

SECONDARY OUTCOMES:
Total operative time. | Intraoperative
  The operation room nurse recorded the time lapse between the skin incision and the end of skin suturing.
The mean estimated intraoperative blood loss. | Intraoperative
  The estimated intraoperative blood loss was evaluated by weighting all surgical sponges, swabs, and drapes before and after use. Using this formula: Blood Loss (mL) = (Wet weight - Dry weight in grams) = mL of blood lost then add this to the volume of blood collected in suction canisters and subtract any irrigation or amniotic fluid.
The number of additional hemostatic sutures needed. | immediately postoperative
  The the obstetrician who performed the procedure recorded this in the participant file.
Uterine niche measurments | At 6 months postpartum
  Using saline-infusion sonohysterography (2 dimensional, sagittal and coronal views). Niche depth, length, width, and residual myometrial thickness are to be recorded.
Menstrual characteristics among participants with uterine niche | At 6 months postpartum
  For participants diagnosed with uterine niche, menstrual history is to obtained by an independent obstetrician/gynecologist, documenting number of spotting days, total bleeding days, amenorrhea, and contraceptive use.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ALNEZAMY, MD, Principal Investigator — Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Locations (1):
- Benha Univesity Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Background] Klein Meuleman SJM, Min N, Hehenkamp WJK, Post Uiterweer ED, Huirne JAF, de Leeuw RA. The definition, diagnosis, and symptoms of the uterine niche - A systematic review. Best Pract Res Clin Obstet Gynaecol. 2023 Aug;90:102390. doi: 10.1016/j.bpobgyn.2023.102390. Epub 2023 Jul 15. PMID 37506497
- [Background] Vervoort A, Vissers J, Hehenkamp W, Brolmann H, Huirne J. The effect of laparoscopic resection of large niches in the uterine caesarean scar on symptoms, ultrasound findings and quality of life: a prospective cohort study. BJOG. 2018 Feb;125(3):317-325. doi: 10.1111/1471-0528.14822. Epub 2017 Aug 28. PMID 28703935
- [Background] Baranov A, Gunnarsson G, Salvesen KA, Isberg PE, Vikhareva O. Assessment of Cesarean hysterotomy scar in non-pregnant women: reliability of transvaginal sonography with and without contrast enhancement. Ultrasound Obstet Gynecol. 2016 Apr;47(4):499-505. doi: 10.1002/uog.14833. Epub 2016 Feb 29. PMID 25720922
- [Result] Osser OV, Jokubkiene L, Valentin L. High prevalence of defects in Cesarean section scars at transvaginal ultrasound examination. Ultrasound Obstet Gynecol. 2009 Jul;34(1):90-7. doi: 10.1002/uog.6395. PMID 19499514
- [Result] Osser OV, Jokubkiene L, Valentin L. Cesarean section scar defects: agreement between transvaginal sonographic findings with and without saline contrast enhancement. Ultrasound Obstet Gynecol. 2010 Jan;35(1):75-83. doi: 10.1002/uog.7496. PMID 20034000
- [Result] Sholapurkar SL. Etiology of Cesarean Uterine Scar Defect (Niche): Detailed Critical Analysis of Hypotheses and Prevention Strategies and Peritoneal Closure Debate. J Clin Med Res. 2018 Mar;10(3):166-173. doi: 10.14740/jocmr3271w. Epub 2018 Jan 26. PMID 29416572
- [Result] Siraj SHM, Lional KM, Tan KH, Wright A. Repair of the myometrial scar defect at repeat caesarean section: a modified surgical technique. BMC Pregnancy Childbirth. 2021 Aug 17;21(1):559. doi: 10.1186/s12884-021-04040-9. PMID 34404382